CLINICAL TRIAL: NCT02841007
Title: gekoTM Neuromuscular Electrostimulation (NMES) Device, Pilot Feasibility Study Looking at Time to Surgery Study in Patients Requiring Ankle Fixation Following Fracture, Comparison to Matched Retrospective Controls
Brief Title: Midds Ankle Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FKD-LOS-001
Record Dates: First submitted 2016-07-15; First posted 2016-07-21 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2016-07

CONDITIONS: Ankle Fracture Requiring Internal Fixation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- geko device arm (Experimental): Patients consenting to take part will receive the geko device prior to surgery to internally fixate their fractured ankle, to reduce and prevent oedema
  Interventions: Device: geko neuromuscular electrostimulation device

INTERVENTIONS:
Device: geko neuromuscular electrostimulation device

SUMMARY:
The geko™ device is indicated for the prevention and treatment of oedema. The aim of this study is to show that recruiting, and performing study assessments in ankle fracture patients requiring surgery to fix their ankle attending the James Cook Hospital is feasible, and to obtain data to support the powering of a larger study to demonstrate the effectiveness of the geko™ device at reducing length of stay for this population of patients. This study will also allow us to assess the acceptability, tolerability and compliance of treatment with the geko device.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years old
2. Clinically and radiologically diagnosed acute ankle fracture that, in the opinion of the treating surgeon, requires operative fixation
3. Able to understand the Patient Information Sheet (PIS) and willing to sign the written Informed Consent Form.
4. Able and willing to follow the protocol requirements.

Exclusion Criteria:

1. Has a pacemaker
2. Morbid Obesity (BMI Index >40kg/m2).
3. Patients who on presentation to hospital are known to be pregnant.
4. Clinically significant co-morbidities that need to be treated prior to surgical intervention and could therefore impact upon time to theatre
5. History or signs of previous deep or superficial vein thrombosis/pulmonary embolism.
6. Varicosities, ulceration or erosion around the area of the leg where the study device would be fitted
7. Diabetic
8. Already taking part in a clinical study, or has so within the last 8 weeks
9. None responder to geko™ device

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Feasibility to recruit n=20 ankle fracture patients in trauma setting within 4 months | 4 months
Time to readiness for surgery | 0-~7days

SECONDARY OUTCOMES:
Oedema reduction in prospective geko™ subjects prior to surgery, by two circumferential measures using tape measures built into the patients plaster cast | 0-~7days
Adverse events, including the need for secondary surgery or additional treatment, serious adverse events | study duration up to ~14days

CONTACTS AND LOCATIONS:
Locations (1):
- James Cook Hospital, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No